CLINICAL TRIAL: NCT01964105
Title: 3D Breast Imaging for Cosmetic and Reconstructive Breast Surgery: Does 3D Improve Patient Reported Outcomes in Primary Breast Augmentation?
Brief Title: 3D Breast Imaging for Cosmetic and Reconstructive Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201210065
Record Dates: First submitted 2013-09-26; First posted 2013-10-17 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Hypomastia; Primary Breast Augmentation
Keywords: Hypomastia; Augmentation; Breast; 3D; Breast Q
MeSH Terms: interventions — Imaging, Three-Dimensional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3D Imaging Simulation (Experimental): Intervention Group: 3D Image Simulation + Standard Preoperative Evaluation Goal: 50 patients
  Interventions: Device: 3D Imaging
- Standard Preoperative Evaluation (No Intervention): Control Group: Patients will receive standard preoperative evaluation (2D imaging).
  Goal: 50 patients
- Non-Randomized Cohort: 3D Imaging (Other): Patients who refuse the option of randomization but otherwise meet the inclusion and exclusion criteria will be offered participation in this study as part of a non-randomized cohort.
  Goal: 50 Patients
  Interventions: Device: 3D Imaging

INTERVENTIONS:
Device: 3D Imaging
  Other Names: Vectra 3D
  Arms: 3D Imaging Simulation; Non-Randomized Cohort: 3D Imaging

SUMMARY:
The purpose of this trial is to evaluate the impact of incorporating three-dimensional (3D)imaging during preoperative consultation on patient reported outcomes in primary breast augmentation surgery. 3D imaging is an innovative technology that allows the surgeon to share with images how one could look after one's procedure. The patient's assessment will be collected using the Breast Q, an objective questionnaire that captures patient satisfaction with breast augmentation.

DETAILED DESCRIPTION:
Consultation for primary breast augmentation involves clear communication between patient and surgeon to select the implant and manage expectations. Tissue-based planning strategies rely on tissue characteristics and measurements to produce safe and reproducible aesthetic outcomes. The implementation of sizers in the preoperative consultation and a greater emphasis on patient aesthetic goals have also proven to be favorable strategies. Recently, many plastic surgeons have started to incorporate three-dimensional (3D) photography and computer simulation into their preoperative consultation process. The accuracy of computer simulation for volume assessment of breast augmentation is reportedly ≥90%, and patients demonstrate a preference for consultations involving simulation.Support for computer simulation, however, is not unanimous.

Quantitative analyses, prospective study designs, and utilization of validated health-related quality of life metrics have been recommended to more thoroughly scrutinize implant selection systems and outcomes in aesthetic surgery.Mammometrics yields numerical data useful for quantifying changes in breast morphology after breast reduction, reconstruction with implants, and augmentation. The BREAST-Q represents the most comprehensive and quantitative method for patient self-assessment following breast surgery, and has gained traction as a patient-reported outcomes instrument for breast augmentation. To date, there are no studies that focus on the impact of simulation on patient-reported outcomes in breast augmentation, as measured with the validated BREAST-Q. Furthermore, there is minimal data examining correlations between patient-reported outcomes and mammometrics.

The purpose of this study was to conduct a prospective, clinical trial to evaluate the impact of 3D imaging and simulation used during the preoperative consultation on postoperative patient-reported outcomes and quantitative changes in breast morphology. We hypothesized that computer simulation would facilitate patient education and surgical planning, thus leading to quantitatively higher patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled for elective breast augmentation cosmetic procedure.

Exclusion Criteria:

* Breast reconstruction for malignancy
* Cognitively unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence M Myckatyn, MD, FACS, Principal Investigator — Washington University School of Medicine
Locations (1):
- West County Plastic Surgeons of Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Tepper OM, Unger JG, Small KH, Feldman D, Kumar N, Choi M, Karp NS. Mammometrics: the standardization of aesthetic and reconstructive breast surgery. Plast Reconstr Surg. 2010 Jan;125(1):393-400. doi: 10.1097/PRS.0b013e3181c4966e. No abstract available. PMID 20048631
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Derived] Overschmidt B, Qureshi AA, Parikh RP, Yan Y, Tenenbaum MM, Myckatyn TM. A Prospective Evaluation of Three-Dimensional Image Simulation: Patient-Reported Outcomes and Mammometrics in Primary Breast Augmentation. Plast Reconstr Surg. 2018 Aug;142(2):133e-144e. doi: 10.1097/PRS.0000000000004601. PMID 30045174
- See also: Click here for Washington University's study location. — http://westcountyplasticsurgeons.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Randomized Cohort: 3D Imaging: Patients who refuse the option of randomization but otherwise meet the inclusion and exclusion criteria will be offered participation in this study as part of a non-randomized cohort.
  Goal: 50 Patients
  3D Imaging
- 3D Imaging Simulation: Intervention Group: 3D Image Simulation + Standard Preoperative Evaluation Goal: 50 patients
  3D Imaging
Period: Overall Study
Arm/Group | Standard Preoperative Evaluation | Non-Randomized Cohort: 3D Imaging | 3D Imaging Simulation
Started | 15 | 75 | 10
Completed | 13 | 62 | 10
Not Completed | 2 | 13 | 0
Not completed — Lost to Follow-up | 2 | 13 | 0

BASELINE CHARACTERISTICS:
Population: All patients presenting for primary breast augmentation that were not excluded. We excluded patients who refused participation in a study, cancelled surgery, had greater than grade I ptosis, congenital deformity of the chest wall, could not commit to 6 months follow-up, needed a concurrent mastopexy, or had concomitant fat transfer to the breast.
Groups:
- 3D Imaging Simulation: The intervention group underwent computer simulation with the Vectra Sculptor package (Canfield Scientific Inc, Parsippany, NJ) in addition to control group preoperative evaluation.
- Standard Preoperative Evaluation: The control group underwent tissue-based planning that was supplemented by review of photos obtained from magazines or the internet, and placement of sizers in a surgical bra. Control group patients underwent three-dimensional photography with the same system but were not simulated.
- Non-Randomized Cohort: 3D Imaging: Since enrollment in the non-randomized arm was predicated upon a pre-existing desire for computer simulation, all of these patients received this intervention.
- Total: Total of all reporting groups
Arm/Group | 3D Imaging Simulation | Standard Preoperative Evaluation | Non-Randomized Cohort: 3D Imaging | Total
Number analyzed (Participants) | 10 | 13 | 62 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (23.1) | 40.2 (11) | 35.8 (8.2) | 37.2 (8.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 10 | 13 | 62 | 85
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 13 | 62 | 85
Volume of Breast [Mean (Standard Deviation); unit: cubic centimeters (cc)] | 494.5 (93) | 503.4 (113.1) | 420 (119.3) | 441 (120.5)
BREAST-Q [Mean (Standard Deviation); unit: units on a scale] — BREAST-Q is a validated measures of patient reported outcomes. For this study we utilized the preoperative and postoperative BREAST -Q designed to analyze outcomes following breast augmentation The BREAST-Q is measured as a Q-score on a scale of 0-100. 0 is a poor score, 100 is an optimal score.
  units on a scale | 63.6 (18.6) | 70.1 (21.5) | 64.8 (19.3) | 64.6 (19.1)

OUTCOME MEASURES:

1. Primary Outcome: Breast Q Augmentation Module
Description: BREAST-Q is a validated measures of patient reported outcomes (this is not an acronym). For this study we utilized the preoperative and postoperative BREAST -Q designed to analyze outcomes following breast augmentation The BREAST-Q is measured as a Q-score on a scale of 0-100. 0 is a poor score, 100 is an optimal score. Q-scores stand independently and are not combined to create a total score.
Time Frame: up to 6 months postop visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard Preoperative Evaluation: Intervention Group: 3D Image Simulation + Standard Preoperative Evaluation Goal: 50 patients
  3D Imaging
- 3D Imaging Simulation: Control Group: Patients will receive standard preoperative evaluation (2D imaging).
  Goal: 50 patients
Arm/Group | Standard Preoperative Evaluation | 3D Imaging Simulation | Non-Randomized Cohort: 3D Imaging
Number analyzed (Participants) | 13 | 10 | 62
units on a scale | 494.5 (93) | 503.4 (113.1) | 420 (119.3)

ADVERSE EVENTS:
Time Frame: 6 months (entire study period)
Description: Adverse events were collected as defined by clinicaltrials.gov
Groups:
- Standard Preoperative Evaluation: Patients undergo standard tissue-based planning. They were randomized to this intervention.
- 3D Imaging Simulation: Patient undergo three-dimensional simulation of their breast augmentation. They were randomized to this intervention.
- Non-Randomized Cohort: 3D Imaging: Patient undergo three-dimensional simulation of their breast augmentation. They sought this intervention (ie. not randomized).
Arm/Group | Standard Preoperative Evaluation | 3D Imaging Simulation | Non-Randomized Cohort: 3D Imaging
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10 | 0/62
Other Adverse Events (participants affected / at risk) | 0/10 | 0/13 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2014-08-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT01964105/Prot_000.pdf
  • Informed Consent Form (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT01964105/ICF_001.pdf
  • Statistical Analysis Plan (2014-08-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT01964105/SAP_002.pdf